CLINICAL TRIAL: NCT02393391
Title: Novel Non Invasive Brain Stimulation Based Treatment for Chronic Low Back
Brief Title: A Novel Non Invasive Brain Stimulation Based Treatment for Chronic Low Back Pain (CLBP)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: NIBS NeuroScience Technologies (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TASMC-14-SB-600-CTIL
Record Dates: First submitted 2015-03-08; First posted 2015-03-19 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NIBS tDCS/tACS stimulation (Active Comparator): Each patient will undergo initial diagnosis with NIBS algorithm utilizing EEG measurements combined with TMS. Initial diagnosis will last 10 minutes in which EEG measurement will be recorded 5 minutes and then in combination with TMS for another 5 minutes with no more than 500 TMS stimuli applied to cortex at low frequency of up to 5Hz. EEG recording will be analyzed by NIBS algorithm which will propose a course of treatment with the following limitations: stimulation of 2mA (32, 33) current after 30 seconds ramp up of 0.1mA increments, 20 min for each session, twice a week
  Interventions: Device: Neuroelectrics STARSTIM
- inactive electrodes (Placebo Comparator): diagnosis and monitoring will be performed as in active treatment, but during treatment anodal/cathodal/alternate stimulation will begin and automatically stop after 30 seconds leaving subject with an inactive electrodes in place for the remainder of treatment duration
  Interventions: Device: Neuroelectrics STARSTIM

INTERVENTIONS:
Device: Neuroelectrics STARSTIM

SUMMARY:
Neuropathic pain results from damage to or dysfunction of the peripheral or central nervous system, rather than stimulation of pain receptors. Diagnosis is suggested by pain out of proportion to tissue injury, dysesthesia (eg, burning, tingling), and signs of nerve injury detected during neurologic examination. Although neuropathic pain responds to opioids, treatment is often with adjuvant drugs (eg, antidepressants, anticonvulsants, baclofen, topical drugs). Neuropathic pain (e.g. phantom limb pain, CRPS, postherpetic neuralgia, postsurgical pain syndromes, CLBP etc.) remains a challenging condition to treat because it is commonly refractory to classical pharmacological and to surgical treatment approaches. Chronic low back pain (CLBP) is a widespread and costly problem for which few interventions are effective. An increased focus on the study of the nervous system and its involvement in pain disorders has documented complex neuronal activity and structural changes at a peripheral, as well as at spinal cord and cortical levels indicating a neuropathic element in CLBP. Accumulated evidence suggests that neuropathic pain in general and CLBP specifically might be associated to brain cortical plastic changes. Thus an ideal rehabilitative approach should aim to reverse them. In line with this idea, the investigators suggest an innovative noninvasive intervention aimed at alleviating neuropathic pain. New rehabilitative approaches have been proposed to try and reverse this cortical reorganization. Results of several studies have shown that motor cortex stimulation with epidural electrodes or repetitive transcranial magnetic stimulation (rTMS) or transcranial direct stimulation (tDCS) are effective in reducing pain in patients with central pain refractory to treatment. Transcranial direct current stimulation (tDCS) is an easily applied and safe technique by which brain activity can be modulated noninvasively and can decrease pain in patients with refractory central pain. The investigators hypothesized that focal-tDCS treatment personally customized to each patients basal neuronal network properties would result in both acute and long term pain relief for neuropathic pain patients.

ELIGIBILITY:
Inclusion Criteria:

1. age 18 to 70
2. CLBP as defined by the European guidelines

Exclusion Criteria:

1. Acute low back pain (duration of less than 6 months
2. Neurological illness causing structural brain damage (e.g. Stroke, TIA)
3. Psychiatric disease other than mood disorders
4. Current chronic use of medications with pro-epileptic properties
5. Known alcohol dependency
6. Use of alcohol within the previous 24 hours
7. History of loss of consciousness
8. Epilepsy or epilepsy in a first degree relative
9. Medical implants
10. Pregnancy
11. Illicit drug use or within the previous month

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-05; Primary Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment efficacy (evaluated by pain level and sleep quality questionnaire) | one year
  Efficacy of the treatment will be evaluated by pain level and sleep quality questionnaire